CLINICAL TRIAL: NCT04245943
Title: Rehabilitation - Physical Activity and Coping
Acronym: RPAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/620
Record Dates: First submitted 2020-01-16; First posted 2020-01-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cancer Survivors
Keywords: Rehabilitation; Physical exercise; Return to work; Fatigue; Cancer survivors
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): 18 weeks supervised strength and aerobic exercise training
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — 18 weeks supervised strength and aerobic exercise training.

SUMMARY:
The project is a non-randomized intervention study with group-based physical exercise. Cancer survivors who have participated in the rehabilitation program at the Center for Education and Rehabilitation are included in the study.

The cancer and cancer treatment have led to patients struggling with physical, mental and social late effects which prevent them from functioning in everyday life and return to work. The purpose of the project is to investigate whether one municipal group training measure can help to lower the threshold for the user to maintain good exercise habits and return to work / everyday life, as well as the effect on the user's physical form and quality of life and the transition between health level and the body itself measure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Women and men
* Regardless of cancer diagnosis
* Resident in Bergen municipality
* Finishes their rehabilitation at The Cancer Center for Education and Rehabilitation spring/summer 2019.

Exclusion Criteria:

* Patients who do not speak or understand Norwegian
* Unable to express themselves in writing
* Unable to perform basic daily tasks
* Display cognitive disorder or severe emotional instability
* Suffer from other debilitating illnesses / conditions that may inhibit physical exercise (heart failure, chronic obstructive pulmonary disease, orthopedic conditions, neurological disorders or the like) will be excluded from the study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Objectively recorded physical activity level | 18 weeks
  Change in objectively recorded physical activity level, measured with the SenseWear ™ Mini Armband (SWA) (BodyMedia Inc. Pittsburgh, PA, USA) as average minutes of moderate- to vigorous intensity physical activity (MVPA) from before intervention to after completion of the intervention.

SECONDARY OUTCOMES:
Change in maximal oxygen uptake measured by VO2max | 18 weeks
  Change in VO2max, measured by a maximal incremental exercise test on a treadmill, from before training intervention to post training intervention.
Change in maximal strength | 18 weeks
  Change in 1 repetition maximum strength in upper and lower body measured from before intervention and after completion of the intervention.
Change in quality of life measured by Short Form Health Survey (SF-36) | 18 weeks
  Change in scores on the Short Form Health Survey (SF-36) from before intervention to after completion of the intervention.
Change in fatigue scores using the Chalder Fatigue Questionaire (FQ) | 18 weeks
  Change in scores on the Chalder Fatigue Questionaire (FQ) from before intervention to after completion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Arving, PhD, Study Director — Helse Bergen, Cancer Center for Education and Rehabilitation
Locations (1):
- Helse Bergen,, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication are to be shared with two master students and their professors/supervisors/researchers who take part in the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available from February 2020 to October 31. 2024